CLINICAL TRIAL: NCT02505490
Title: The Effect of Television Watching on Liking of Food in Normal Weight Adults 18-35
Brief Title: The Effect of Television Watching on Liking of Food
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Tennessee, Knoxville (Other)
Responsible Party: Principal Investigator, Hollie Raynor, Professor, The University of Tennessee, Knoxville
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Other
Other Study IDs: UTK IRB-15-02352-XP
Record Dates: First submitted 2015-07-06; First posted 2015-07-22 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Hunger
Keywords: Lunch; Television; Macaroni and Cheese; Salad tossed in dressing
MeSH Terms: interventions — Television

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- No Television (Experimental): The purpose is to determine whether a change in liking of food will occur with a lack of television.
  Interventions: Other: No Television
- Television (Experimental): The purpose is to determine whether a change in liking of food will occur while watching television.
  Interventions: Other: Television

INTERVENTIONS:
Other: Television — The purpose is to determine whether television impacts liking of food.
  Arms: Television
Other: No Television — The purpose is to determine whether the lack of television impacts liking of food.
  Arms: No Television

SUMMARY:
The purpose of the study is to investigate the effect of television viewing on liking of food.

DETAILED DESCRIPTION:
The objective of this investigation is to determine whether participants will have a change of liking of food based on television viewing. The specific aims of the study are:

1. Determine the effect of television on liking of food.
2. Determine the effect of no television on liking of food.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 35 years
* Body mass index (BMI) between 18.5 kg/m2 and 24.9 kg/m2
* Unrestrained eater (≤ 12 on the Three Factor Eating Questionnaire [TFEQ-R])
* Report a favorable preference for foods served in the meal including: macaroni and cheese and salad (dressing will be chosen by the participant via initial phone screen), participants must rate each food item ≥ 3 during phone screen and ≥ 50 on a visual analogue scale (VAS) during the initial screening session
* Regularly eat a meal before 10:00 am
* Are able to complete all sessions within eight weeks of the screening session
* Report being a non-smoker
* Are not taking medications that affect appetite or food intake
* Are not pregnant or breastfeeding
* Are not on a dietary plan or have dietary restrictions that prevent consumption of certain types and/or amounts of food

Exclusion Criteria:

* Binge eating; and/or
* Athletes in training

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
The Effect of Television Watching on Liking of Food via Visual Analog Scale | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Rosenthal, BS, Principal Investigator — The University of Tennessee, Knoxville
Locations (1):
- University of Tennessee, Knoxville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided